CLINICAL TRIAL: NCT02333786
Title: Comparison of Long-axis/In-plane and Short-axis/Out-of-plane Methods During the Ultrasound-guided Arterial Cannulation in Pediatric Patients
Brief Title: Ultrasound-guided Arterial Catheterization in Pediatric Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jin-Tae Kim, Assistant professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: H-1409-095-610
Record Dates: First submitted 2015-01-05; First posted 2015-01-07 (Estimated); Last update posted 2015-10-07 (Estimated); Status verified 2015-10

CONDITIONS: Ultrasound; Arterial Catheterization; Child

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Infant (Experimental): Radial artery or posterior tibial artery of patients younger than 1 year old are either cannulated with short-axis/out-of-plane or long-axis/in-plane US-guided arterial catheterization technique.
  Interventions: Other: Long-axis/in-plane US-guided arterial catheterization; Other: Short-axis/out-of-plane US-guided arterial catheterization
- Preschool child (Experimental): Radial artery or posterior tibial artery of patients older than 1 year old and younger than 5 years old are either cannulated with long-axis/in-plane or short-axis/out-of-plane US-guided arterial catheterization technique.
  Interventions: Other: Long-axis/in-plane US-guided arterial catheterization; Other: Short-axis/out-of-plane US-guided arterial catheterization

INTERVENTIONS:
Other: Long-axis/in-plane US-guided arterial catheterization — Cannulate the radial artery or posterior tibial artery of an infant of a preschool child putting the 24 gauge needle parallel to the ultrasound transducer.
Other: Short-axis/out-of-plane US-guided arterial catheterization — Cannulate the radial artery or posterior tibial artery of an infant or a preschool child putting the 24 gauge needle perpendicular to the ultrasound transducer.

SUMMARY:
Investigators designed a prospective randomized controlled study to compare the long-axis/in-plane and short-axis/out-of-plane methods during the ultrasound-guided arterial catheterization in pediatric patients younger than 5 years old.

ELIGIBILITY:
Inclusion Criteria:

* Surgery under general anesthesia
* Requires invasive arterial blood pressure monitoring

Exclusion Criteria:

* Infection/hematoma/skin disease/arteriovenous fistula/recent catheterization scar in radial artery or posterior tibial artery
* Peripheral vascular disease
* Congenital aortic disease

Max Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 108 (Actual)
Dates: Start 2015-01; Primary Completion 2015-04 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Arterial catheterization time | Interval between contact of the ultrasound transducer with the skin and confirmation of an arterial waveform on the monitor, an expected average of 200 seconds

SECONDARY OUTCOMES:
Ultrasound imaging time | Interval between contact of the ultrasound transducer with the skin and penetration of the needle through the skin, an expected average of 30 seconds
Time to first puncture of the artery | Interval between skin penetration of the needle and flashback of blood, an expected average of 100 seconds
Number of puncture attempts | Up to 5 times, an expected average observation time of 600 seconds

CONTACTS AND LOCATIONS:
Overall Officials: Jin-Tae Kim, MD. PhD., Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, Seoul, South Korea

REFERENCES:
- [Derived] Song IK, Choi JY, Lee JH, Kim EH, Kim HJ, Kim HS, Kim JT. Short-axis/out-of-plane or long-axis/in-plane ultrasound-guided arterial cannulation in children: A randomised controlled trial. Eur J Anaesthesiol. 2016 Jul;33(7):522-7. doi: 10.1097/EJA.0000000000000453. PMID 26986774